CLINICAL TRIAL: NCT07177144
Title: Does Vnotes Salpingectomy Reduce Ovarian Reserve?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Yıldız, associate professor of gynecology and obstetrics, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Gaziosmanpasatrehmh
Record Dates: First submitted 2025-08-18; First posted 2025-09-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Vnotes; Salpingectomy; Ovarian Reserve
Keywords: vnotes; salpingectomy; ovarian reserve
MeSH Terms: interventions — Anti-Mullerian Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vnotes salpingectomy performed (Experimental): group of women who underwent salpingectomy with the vnotes method for women who wanted to have their tubes removed for contraception
  Interventions: Other: anti müllerian hormone; Diagnostic Test: anti müllerian hormon
- laparoscopic salpingectomy performed (Active Comparator): group of women who underwent salpingectomy with the laparoscopic salpingectomy method for women who wanted to have their tubes removed for contraception
  Interventions: Other: anti müllerian hormone; Diagnostic Test: anti müllerian hormon

INTERVENTIONS:
Other: anti müllerian hormone — participants were checked for amh levels preoperatively
Diagnostic Test: anti müllerian hormon — participants were checked for amh levels at 3 months postoperatively.

SUMMARY:
Comparison of Transvaginal Natural Orifice Transluminal Endoscopic Surgery and Conventional Laparoscopy in terms of their effects on ovarian reserve in Opportunistic Bilateral Salpingectomy for Permanent Female Sterilization

DETAILED DESCRIPTION:
The study will include participants who apply to our clinic for salpingectomy for contraception and agree to participate in the study. vnotes salpingectomy method or classical laparoscopic salpingectomy will be offered to the patients as two salpingectomy methods and the patient will be included in whichever group in the study. All surgeries will be performed by the same surgeon. 3 months after the date of surgery, the patient will be called for a follow-up for amh repeat and the two groups will be compared both within themselves and with each other to evaluate whether the different surgical technique has an effect on ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* to want to have your tubes removed, not to have undergone tubal and ovarian surgery before, not to use hormones and medications that can affect the level of sex hormones and its levels,

Exclusion Criteria:

* not being in the specified age range (18-45), having a history of tubal ligation, having tubal cancer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
measuring anti-millerian hormone level | amh level (ng/ml) will be checked before the operation, and after 3 months, she will be called for control and measured again.
  To evaluate the effect of two surgical methods on ovarian reserve by measuring serum anti-Müllerian hormone levels (ng/ml) before surgery and after salpingectomy.

SECONDARY OUTCOMES:
comparison of duration of surgery | Perioperative
  To compare the success of the two surgical techniques Surgery duration: the time from when the patient first receives anesthesia until they are awakened, recorded in minutes (min)
Postoperative hospital stay duration | Perioperative
  The days the patient stays in the hospital, starting from the first day they are admitted for surgery until they are discharged after full recovery following the surgery, will be recorded as days. the number of days the patient stays in the hospital, recorded in days (days)
postoperative pain | first hour after surgery
  The patient is asked to rate the pain they feel from the moment they wake up after surgery on a scale of 1 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The name, surname and personal data of the patients will never be shared with anyone. Data related to the study such as surgical information, amh level, antral follicle count, etc. specified in the informed consent obtained for the study will be used.

REFERENCES:
- [Result] Yassa M, Kaya C, Kalafat E, Tekin AB, Karakas S, Mutlu MA, Birol P, Tug N. The Comparison of Transvaginal Natural Orifice Transluminal Endoscopic Surgery and Conventional Laparoscopy in Opportunistic Bilateral Salpingectomy for Permanent Female Sterilization. J Minim Invasive Gynecol. 2022 Feb;29(2):257-264.e1. doi: 10.1016/j.jmig.2021.08.009. Epub 2021 Aug 16. PMID 34411729
- [Derived] Yildiz E, Coskun ES, Timur GY, Bacak HB, Aciyiyen Y, Terkan H, Bilici SR, Ersoy D, Aldanmaz B, Salman S. When performing vNOTES salpingectomy, are we damaging the ovarian reserve? Results from a randomized, controlled trial. J Minim Invasive Gynecol. 2026 Feb 7:S1553-4650(26)00103-2. doi: 10.1016/j.jmig.2026.02.009. Online ahead of print. PMID 41662907